CLINICAL TRIAL: NCT04185714
Title: THE EFFECTS OF KINESIO®TAPING ON PAIN, DISABILITY AND QUALITY OF LIFE IN PATIENTS WITH MIGRAINE: A RANDOMISED SINGLE-BLIND, PLACEBO-CONTROLLED TRIAL
Brief Title: THE EFFECTS OF KINESIO®TAPING IN PATIENTS WITH MIGRAINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Esra Kınacı, Research Asistant, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098-604.01.1
Record Dates: First submitted 2019-11-25; First posted 2019-12-04 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Migraine; Pain
Keywords: Episodic Migraine; Kinesiotape; Pain; Physiotherapy; Disability; Pressure Pain Threshold; Quality of Life
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Experimental group will be applied Kinesotaping , exercise programme will be given.
  Interventions: Other: Kinesiotaping
- Control group (No Intervention): Exercise programme will be given.
- Placebo group (Placebo Comparator): Sham taping will be applied, exercise programme will be given.
  Interventions: Other: Placebo taping

INTERVENTIONS:
Other: Kinesiotaping — Kinesiotaping (KT) is an approach that supports injured muscles and joints and helps relieve pain.
  Other Names: exercise; sham taping
  Arms: Experimental group
Other: Placebo taping — sham taping
  Arms: Placebo group

SUMMARY:
In patients with migraine, neck pain and trigger points in the neck muscles are common in clinical practice. This study was to investigate whether kinesiotaping applied to the cervical muscles has a clinical effect on pressure pain threshold, disability and quality of life in patients with migraine.

DETAILED DESCRIPTION:
Patients with episodic migraine who were followed up by department of neurology in regional hospital will be included in the study. The Clinical Research Ethics committee approved the study (protocol no 10840098-604.01.1-E.6803).

Inclusion criterias are aged between 18-55 years, the patients with episodic migraine by neurologist according to ICHD-3 Beta criteria, patients with episodic migraine and associated neck pain, headache frequency in 1 month < 15 days and pain severity according to VAS above 40 mm.

Exclusion criterias are other headache types, contraindication for KT technique, cervical disc disorders, systemic rheumatic disease, fibromyalgia pain syndrome, myofascial pain syndrome, temporamandibular joint dysfunction, pregnancy, overuse medication, patients who had gotten rehabilitation programme before at least 3 months ago and anaesthetic blockage before at least 6 months ago.

All patients will allocate three groups. The patients with episodic migraine were randomly assigned to control group (n=20), placebo group (n=20) and experimental group (n= 20).

Outcome measures Demographic data and headache characteristics of the patients (frequency, duration, onset of headache, family history, onset age of headache, pain triggering factors, and localization of headache), presence of neck pain and disability of the last 1 month will evaluate before and after 6 weeks of treatment via self-administered questionnaire. Pressure Pain Algometry (Baseline Dolorimeter), Visual Analogue Scale (VAS), Neck Disability Index, Migraine Disability Assessment Scale (MIDAS) and Short Form-36 (SF-36) will use as the assessment method in the 6-week follow-up.

Intervention All two groups will give a 6-week exercise programme for 2 days per week. Exercise programme that included neck and head isotonic and isometric exercises show by physiotherapist. The participants will administer the exercises every day for 45 minutes. Sham taping will be applied for the placebo group. Kinesiotaping will be applied to the trapezius and deep cervical muscles twice a week for experimental group. The taping replace every 3 days.

Statistical Analyses Data will be expressed as mean, standard deviation and median. Significance between pre- and post-treatment pain, disability and quality of life variables was statistically significant with Paired Stutend's t - test and Wilcoxon signed rank tests; The differences between groups will be analysed using the Kruskal-Wallis-test to determine statistical significance. For statistical significance p <0.05 probability value will be accepted.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria

* age between 18-55 years,
* the patients with episodic migraine by neurologist according to ICHD-3 Beta criteria,
* headache frequency in 1 month < 15 days and
* pain severity according to VAS above 40 mm.

Exclusion Criteria:

* other headache disorders
* disc disorders,
* systemic rheumatic disease, fibromyalgia pain syndrome, myofascial pain syndrome,
* temporamandibular joint dysfunction,
* pregnancy,
* overuse medication,
* patients who had gotten rehabilitation programme before at least 3 months ago and
* anaesthetic blockage before at least 6 months ago.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
visual analog scale | Pretreatment- Posttreatment ( 6 weeks later)
  Headache pain severity
visual analog scale | Pretreatment-Posttreatment (6 weeks later)
  Neck pain severity
Baseline Dolorimeter | pretreatment- Posttreatment ( 6 weeks later)
  pressure pain threshold
Clinical data questionnaire | pretreatment- Posttreatment ( 6 weeks later)
  clinical data

SECONDARY OUTCOMES:
Short form-36 | pretreatment - Post treatment (6 weeks later)
  quality of life
MIDAS | Pretreatment
  Migraine Disability Assessment Scale (not score scale It describes the total of 3-month headache )
Neck Disability Index | pretreatment - Post treatment (6 weeks later)
  questionnaire to assess neck pain related disability

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biber EK, Polat B. Effects of kinesiotaping combined with physical therapy in patients with migraine-associated neck pain: a randomized controlled study. BMC Musculoskelet Disord. 2025 Oct 23;26(1):990. doi: 10.1186/s12891-025-08985-2. PMID 41131499